CLINICAL TRIAL: NCT01397253
Title: Virtual Continuity and Its Impact on Complex Hospitalized Patients' Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 3130920
Record Dates: First submitted 2011-07-15; First posted 2011-07-19 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-03

CONDITIONS: Automated Communication Tools; Complex Medical Patients
Keywords: Automated Communication Tools; Medication errors; PCP communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- (Usual) MedTrak system of PCP notification (No Intervention): MedTrak, the information system used by the University of Pittsburgh Medical Center (UPMC), currently notifies PCPs when patients are admitted and discharged from the hospital.
- Automated communication tools (Experimental): An enhanced version of MedTrak (the present system of PCP notification). Electronic medical record links will be developed and used to allow automated communication with the PCP.
  Interventions: Other: Automated communication tools

INTERVENTIONS:
Other: Automated communication tools — Automated communication tools will include:
  * PCP notification of patient admission and location
  * Data on medications begun on admission
  * Automated alerts on changes in patient status and location while the patient is hospitalized
  * Links to the EMR and to hospital physician contact information on all email alerts
  * Real-time delivery of discharge information (medications, instructions, and follow-up) to the PCP
  * Automatic reporting to PCPs of test results pending at discharge
  * Electronic delivery of final discharge summaries
  Arms: Automated communication tools

SUMMARY:
Communication between physicians caring for a patient in the hospital and that patient's primary care provider is less than optimal, and can lead to diminished health care quality and safety. This project will lead to better communication between physicians and could decrease medication errors that tend to occur as the patient goes from hospital to home.

DETAILED DESCRIPTION:
Communication between physicians caring for hospitalized patients and those patients' primary care providers (PCPs) is often suboptimal. Hospital-based information systems can improve communication by automating information exchange between hospital physicians and PCPs, and perhaps, as a result, improve the quality and safety of health care. MedTrak, the University of Pittsburgh Medical Center (UPMC) electronic physician communication tool, has proven successful and is poised to move forward with an initiative the investigators call virtual continuity, allowing PCPs to follow their patients electronically if they cannot do so physically. Virtual continuity will include: emails to PCPs triggered by clinical events with embedded links to electronic medical record data and communication portals, medication lists electronically delivered to PCPs at admission and discharge, and immediate PCP notification of discharge with pertinent clinical details. To evaluate virtual continuity, the investigators will examine the frequency of discharge medication errors in complex medical patients using a pre-post study design of virtual continuity compared to usual communication. Medication errors will be ascertained using accepted methods. The investigators will also investigate differences in rehospitalization, post discharge emergency department visit and PCP follow up rates. The IT cost of implementing and maintaining the virtual continuity intervention will also be assessed. Virtual continuity will allow PCPs to participate more directly in the care of their hospitalized patients. Improved communication could lead to higher-quality patient care and greater patient care safety for hospitalized patients with complex medical problems.

ELIGIBILITY:
Inclusion Criteria:

* Are admitted to UPMC Presbyterian General Medicine, Geriatrics, Cardiology, or Surgery inpatient services;
* Are 18 years of age or older;
* Are currently receiving 5 or more medications;
* Have 2 or more comorbid conditions present, defined using the Elixhauser comorbidity system (Med Care 1998;36:8-27 and Med Care. 2005 Nov; 43(11): 1130-9 ). These comorbidities are: congestive heart failure, cardiac arrhythmias, valvular disease, pulmonary circulation disorders, peripheral vascular disorders, hypertension, paralysis, other neurologic disorders, chronic pulmonary disease, diabetes uncomplicated, diabetes complicated, hypothyroidism, renal failure, liver disease, peptic ulcer disease excluding bleeding, AIDS/HIV disease, lymphoma, metastatic cancer, solid tumor without metastasis, rheumatoid arthritis/collagen vascular diseases, coagulopathy, obesity, weight loss, fluid and electrolyte disorders, blood loss anemia, deficiency anemias, alcohol abuse, drug abuse, psychoses, and depression
* Have a Primary Care Physician who has outpatient data included on EPIC electronic health record.

Exclusion Criteria:

* Are admitted to critical care units;
* Are admitted from skilled nursing facilities;
* Have dementia;
* Were previously enrolled in the study
* Are organ transplant recipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2010-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Smith, MD, MS, Principal Investigator — University of Pittsburgh Medical Center, University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Halasyamani L, Kripalani S, Coleman E, Schnipper J, van Walraven C, Nagamine J, Torcson P, Bookwalter T, Budnitz T, Manning D. Transition of care for hospitalized elderly patients--development of a discharge checklist for hospitalists. J Hosp Med. 2006 Nov;1(6):354-60. doi: 10.1002/jhm.129. PMID 17219528
- [Background] Kripalani S, Jackson AT, Schnipper JL, Coleman EA. Promoting effective transitions of care at hospital discharge: a review of key issues for hospitalists. J Hosp Med. 2007 Sep;2(5):314-23. doi: 10.1002/jhm.228. PMID 17935242
- [Background] Kripalani S, LeFevre F, Phillips CO, Williams MV, Basaviah P, Baker DW. Deficits in communication and information transfer between hospital-based and primary care physicians: implications for patient safety and continuity of care. JAMA. 2007 Feb 28;297(8):831-41. doi: 10.1001/jama.297.8.831. PMID 17327525
- [Background] Coleman EA, Boult C; American Geriatrics Society Health Care Systems Committee. Improving the quality of transitional care for persons with complex care needs. J Am Geriatr Soc. 2003 Apr;51(4):556-7. doi: 10.1046/j.1532-5415.2003.51186.x. No abstract available. PMID 12657079
- [Background] Coleman EA, Mahoney E, Parry C. Assessing the quality of preparation for posthospital care from the patient's perspective: the care transitions measure. Med Care. 2005 Mar;43(3):246-55. doi: 10.1097/00005650-200503000-00007. PMID 15725981

RESULTS

PARTICIPANT FLOW:
Groups:
- Automated Communication Tools: An enhanced version of MedTrak (the present system of PCP notification). Electronic medical record links will be developed and used to allow automated communication with the PCP.
  Automated communication tools will include:
  * PCP notification of patient admission and location
  * Data on medications begun on admission
  * Automated alerts on changes in patient status and location while the patient is hospitalized
  * Links to the EMR and to hospital physician contact information on all email alerts
  * Real-time delivery of discharge information (medications, instructions, and follow-up) to the PCP
  * Automatic reporting to PCPs of test results pending at discharge
  * Electronic delivery of final discharge summaries
Period: Overall Study
Arm/Group | (Usual) MedTrak System of PCP Notification | Automated Communication Tools
Started | 443 | 392
Completed | 317 (Primary analysis, remaining patients included in a sensitivity analysis) | 243 (Primary analysis, remaining patients included in a sensitivity analysis)
Not Completed | 126 | 149
Not completed — Reviewed by only 1 pharmacist | 126 | 149

BASELINE CHARACTERISTICS:
Population: Hospitalized medical patients with ≥2 comorbidities and ≥5 chronic medications, at a single center
Groups:
- Total: Total of all reporting groups
Arm/Group | (Usual) MedTrak System of PCP Notification | Automated Communication Tools | Total
Number analyzed (Participants) | 317 | 243 | 560
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 63 [53 to 76] | 63 [54 to 73] | 63 [54 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 150 | 328
  Male | 139 | 93 | 232
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 316 | 242 | 558
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 96 | 86 | 182
  White | 216 | 151 | 367
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 317 | 243 | 560

OUTCOME MEASURES:

1. Primary Outcome: Medication Errors at Hospital Discharge
Description: Medication name, dose, and frequency of administration for patient pre-admission medications will be recorded. Medications received during the hospitalization and discharge medications will be obtained by medical record review following hospital discharge. Pre-admission medications will be compared to discharge medications and differences will be considered discharge medication variances. Two trained pharmacists will independently review medication variances to determine clinical indications or medication errors.
Time Frame: Approximately 1-30 days
Population: Hospitalized medical patients with ≥2 comorbidities and ≥5 chronic medications, at a single center
Measure: Number; unit: Errors
Units Other Than Participants: Number of medications
Arm/Group | (Usual) MedTrak System of PCP Notification | Automated Communication Tools
Number analyzed (Participants) | 317 | 243
Number analyzed (Number of medications) | 3490 | 2823
Errors | 645 | 359

2. Secondary Outcome: Patient PCP Visits, Emergency Room Visits and Rehospitalizations Within 30 Days Post-discharge.
Description: Details regarding patient PCP follow-up office appointments, ER visits and rehospitalizations occuring within 30 days post-discharge will be collected from the EMR.
Time Frame: Within 30 post-discharge from hospital
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | (Usual) MedTrak System of PCP Notification | Automated Communication Tools
Serious Adverse Events (participants affected / at risk) | 0/317 | 0/243
Other Adverse Events (participants affected / at risk) | 0/317 | 0/243

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No